CLINICAL TRIAL: NCT06558565
Title: Efficacy of Stromal Vascular Fraction Versus Platelet Rich Plasma in Treatment of Androgenitic Alopecia:Randomized Clinical Trial
Brief Title: Efficacy of Stromal Vascular Fraction Versus Platelet Rich Plasma in Treatment of Androgenitic Alopecia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Asmaa Sobhy Afifi Mohamed Aamer, dermatology resident, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-260-2023
Record Dates: First submitted 2024-02-18; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Androgenetic Alopecia
Keywords: stromal vascular fraction - PRP- androgenetic alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: each patient will receive single session of SVF in one half of the frontal scalp & single session of PRP in the other half of the scalp to compare the effectiveness of them in AGA treatment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stromal vascular fraction side (Active Comparator): stromal vascular fraction will be injected in one half of the frontal scalp
  Interventions: Procedure: stromal vascular fraction or platelet rich plasma
- PRP side (Active Comparator): PRP will be injected in the other half of frontal scalp
  Interventions: Procedure: stromal vascular fraction or platelet rich plasma

INTERVENTIONS:
Procedure: stromal vascular fraction or platelet rich plasma — stromal vascular fraction will be injected in one half of the scalp & PRP will be injected in the other half

SUMMARY:
The goal of this randomized controlled clinical trial is to test the efficacy & safety of stromal vascular fraction in treatment of AGA & compare it to PRP The main questions it aims to answer are:

* efficacy & safety of SVF for treatment of AGA patients
* comparing it to PRP in treatment of AGA Participants will receive a single session of SVF in one half of the scalp & a single session of PRP in the other half.

DETAILED DESCRIPTION:
* History taking from the patients is done about age, duration of the disease previous treatment, medical, surgical history & family history.
* Patients are subjected to clinical evaluation of severity using Hamilton classification & photographing of the patients. In addition, tricoscopic evaluation of hair density & thickness.
* Randomization of patients: The side assigned to SVF treatment is randomized by closed envelop technique.
* Isolation of SVF:

After choosing the site of aspiration (either the hip or the abdomen), sterilization of the site is done.Then, local anesthesia (1 ml of lidocaine 2%) is injected intradermally, small incision (3 ml) is made using sterile blade for insertion of the canula. After that, the tumescence is created with a multiperforated blunt cannula injecting the tumescent solution (0.05% lidocaine in saline solution &1: 200000 epinephrine) then we wait for 20 minutes, followed by harvesting of 50 ml of fat using 2.4 mm microport harvester cannulas with barbed & beveled 1 mm ports. Processing of fat is started by washing of obtained fat using ringer lactate which is left for 10 minutes to decant & elements in the lowest layer is discarded. After that, fat is passed 30 times between two Luer lock 20-ml syringes connected to each other by connectors 2.4mm, 1.4mm, and 1.2mm arranged from higher diameter to lower diameter with minimal pressure force in order to achieve successful mechanical micronization of fat. Then, centrifugation of the micronized fat is done (2000 g for 15 minutes). As a result of this process, 3 layers (oil, fat & SVF) are obtained depending on the density with the SVF pellet suspended in the bottom. After isolation of SVF in one -ml syringes (4-5ml), the scalp is injected with 0.1 ml/cm2 of SVF intra-dermally with small 30 G needle.

- Isolation of platelet-rich plasma: Under sterilized conditions, 8 cc of whole blood are withdrawn from the antecubital vein of each patient. Blood is taken in commercially available PRP kit (Tray Life Tube Gel) containing preformed gel comprising a mixture of polymers that separated plasma, and sodium citrate solution which acts as an anticoagulant. And then is centrifuged at 650 g for 10 minutes. After centrifugation, red blood cells are trapped under the gel, and the upper 1 mL of platelet-poor plasma is removed, and 5 mL PRP obtained.

* Injection of stromal vascular fraction and platelet-rich plasma: Scalp of every patient is divided into two equal halves by the median plane (split scalp), leaving 1.5 cm on both sides of the median plane to minimize diffusion of the injected material to the other side, Lignocaine gel is applied on scalp of patients half an hour before injection followed by sterilization of the site of injection. Then, SVF is injected in one half of scalp & PRP is injected in the other half of scalp, Intra-dermal injections are given by using insulin syringes at 0.1 ml/cm2 interval. Each patient undergoes one session of injection and is followed up for 6 months after the last session.
* Assessment Three & six months After PRP and SVF therapy, the improvement is assessed using pre- and post-treatment photographs according to Hamilton Norwood scale, patient global assessment (PaGAS) scores, physician global assessment (PhGAS) scores, patient satisfaction score, pull test & tricoscopic assessment of:The trichoscopic features of the four areas (bilateral frontal & occipital areas) which are received and analyzed using the trichoscale analysis system of the fotofinder in an area of approximately 1cm2 (0.903 cm2) e.g.hair density & thickness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Hamilton score I to VI in male patients.

Exclusion Criteria:

* Patients with active infection, malignancy, autoimmune disease, and on current anticoagulant therapy.
* Patient on chemotherapy during the last 5 years.
* patients on topical or systemic treatment of AGA

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
comparison of SVF versus PRP | at 3 & 6 months after the sessions
  to compare the mean difference in hair density,thickness, Norwood Hamilton scale, patient global assessment, patient satisfaction & physician global assessment scores between SVF & PRP.

SECONDARY OUTCOMES:
Detecting efficacy of SVF in treatment of AGA | at 3 & 6 months
  To detect provment in hair thickness & diameter

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No